CLINICAL TRIAL: NCT00207428
Title: Randomized, Placebo Controlled, Double Blind Study of Carbamazepine in Treatment of Bronchial Asthma
Brief Title: Antiepileptic Drug Carbamazepine in Treatment of Bronchial Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre of Chinese Medicine, Georgia (Other)
Collaborators: Rea Rehabilitation Centre, Georgia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LP-CZ-0999-0400
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2006-05-16 (Estimated); Status verified 1999-07

CONDITIONS: Bronchial Asthma
Keywords: Bronchial asthma; Carbamazepine; Efficacy
MeSH Terms: conditions — Asthma | interventions — Carbamazepine

INTERVENTIONS:
Drug: Carbamazepine

SUMMARY:
The purpose of this study was evaluation the efficacy of antiepileptic drug carbamazepine in the treatment of mild-to-severe bronchial asthma.

DETAILED DESCRIPTION:
Effective therapy of asthma still remains quite serious problem. According current opinion of leading specialists, asthma is an inflammatory disorder. But asthma also is a paroxysmal disorder: many specialists underline paroxysmal clinical picture of asthma. According to some authors, neurogenic inflammation may play important role in asthma mechanism. But migraine and trigeminal neuralgia are also neurogenic inflammatory paroxysmal diseases, and some antiepileptic drugs, like carbamazepine and valproates, are very effective in therapy of these diseases - more than in 80% of cases. If bronchial asthma also is paroxysmal inflammatory disease, we can suppose a possibility that some antiepileptic drugs also may show high efficacy in asthma therapy. Taken in consideration this hypothesis, we performed a double-blind, placebo-controlled 3-month trial for evaluation of carbamazepine efficacy in treatment of patients with mild-to-severe bronchial asthma.

Comparison: Patients received investigational drug in addition to their usual routine antiasthmatic treatment, compared to patients received placebo in addition to their usual routine antiasthmatic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Out patients
* Bronchial asthma has been known at least for 1 year
* Absence of long-term remissions of asthma (lasting more than 1 month)
* Poorly controlled asthma, due to various reasons
* Non-smokers

Exclusion Criteria:

* Presence of concomitant acute or chronic severe diseases
* Abnormal baseline haematology, blood chemistry or urinalysis
* Allergy or adverse reactions to investigational drug
* Age younger than 16 years old
* Long-term history of smoking
* Pregnancy or lactating

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65
Dates: Start 1999-08; Study Completion 2000-04

PRIMARY OUTCOMES:
At 3 months of treatment: Change from baseline of the PEFR (also %predicted); Number of patients without asthma symptoms

SECONDARY OUTCOMES:
At 3 months of treatment: PEFR before and after salbutamol inhalation;
Difference in PEFR pm-am (in %); The daily (daytime and night-time) symptoms scores; Use of other antiasthmatic medication

CONTACTS AND LOCATIONS:
Overall Officials: Merab Lomia, MD, PhD, Principal Investigator — "Rea" Rehabilitation Centre; Manana Tchaia, MD, Study Director — Centre of Chinese Medicine

REFERENCES:
- See also: Website of Neuroasthma Group — http://www.asthma.ge